CLINICAL TRIAL: NCT03025685
Title: "TransRadial Ultra Support Technique" (TRUST Technique) Versus Anchoring Technique to Enhance Guiding Catheter Support: a Prospective Randomized Pilot Study
Brief Title: "TransRadial Ultra Support Technique" (TRUST)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRUST
Record Dates: First submitted 2017-01-12; First posted 2017-01-19 (Estimated); Last update posted 2017-12-27 (Actual); Status verified 2017-12

CONDITIONS: Coronary Arterioscleroses; Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Coronary Artery Disease; Wire; Coronary stenting
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRUST technique + Coronary Stenting (Experimental): PCI with coronary stenting using TransRadial Ultra Support technique for support improvement
  Interventions: Procedure: TRUST technique; Procedure: Coronary stenting
- Anchoring technique + Coronary Stenting (Active Comparator): PCI with coronary stenting using Wire Anchoring Pass technique for support improvement
  Interventions: Procedure: Anchoring Technique; Procedure: Coronary stenting

INTERVENTIONS:
Procedure: TRUST technique — A soft hydrophilic wire easily pass through the invisible small vessels in the distal parts of a coronary artery into a heart cavity. It is necessary to pass a wire softly and forward as deep as possible. Quite often the wire goes through the left ventricle to aorta arch, and sometimes distal soft tip can be visible in a descending aorta. Thus the stiffest part of the wire become staying on all length of artery, straightening bends and giving the maximum support. After that balloons and stents can be delivered more easily
  Arms: TRUST technique + Coronary Stenting
Procedure: Anchoring Technique — A standard endovascular technique of coronary wire support improvement
  Arms: Anchoring technique + Coronary Stenting
Procedure: Coronary stenting — A standard endovascular procedure of percutaneous coronary intervention with coronary stenting

SUMMARY:
Adequate support is required for challenging percutaneous coronary interventions (PCI). The "TransRadial Ultra Support Technique" (TRUST technique) is a new support technique that provides active support by deep pass of the coronary wire into the heart cavities (left ventricle-LV, right ventricle-RV) or aorta.

ELIGIBILITY:
Inclusion Criteria:

* Subjects singed informed consent form
* Subjects eligible for percutaneous coronary intervention

Exclusion Criteria:

* Age <18 years or >75 years
* Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3.
* Known non-adherence to double anti-platelet therapy (DAPT)
* LVEF <30%
* Continuing bleeding
* Acute coronary syndrome (ST-elevation Myocardial infarction)
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Procedural success | 1 week after PCI
  Device success without the occurrence of in-hospital MACCE
Device success | Intraoperative
  Achievement of a final residual diameter stenosis <20% and a TIMI 3 flow in the target vessel

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No